CLINICAL TRIAL: NCT04456387
Title: An Open-Label, Multicenter Evaluation of the Safety and Efficacy of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection (FRSW107) in Adolescent and Adult Patients With Hemophilia A.
Brief Title: An Open Label Study to Determine the Safety and Efficacy of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection in Adolescent and Adult Patients With Hemophilia A.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhengzhou Gensciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTR20201212
Record Dates: First submitted 2020-06-22; First posted 2020-07-02 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2020-10

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Efficacy and Safety; Factor VIII-Fc Fusion Protein; Adolescent and Adult Patients; Phase III; Pharmacokinetics
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1-on demand treatment (Experimental): Part A-Participants will receive on-demand treatment with Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection for 6 months.
  Interventions: Drug: Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection
- Arm 2- prophylaxis treatment (Experimental): Part B-Participants will receive prophylaxis treatment with Recombinant Human Coagulation Factor VIII-Fc fusion for 6 months.
  12 Participants of them will receive PK assessment at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.)，measured by one-stage assay, they would not be given prophylaxis treatment until the completion of PK blood collection.
  Interventions: Drug: Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection

INTERVENTIONS:
Drug: Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection — Participants received on-demand treatment, doses range from 30 IU/kg to 50 IU/kg, or doses divided on the discretion of the Investigator.
  Arms: Arm 1-on demand treatment
Drug: Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection — Participants received prophylaxis treatment at 50 IU/kg every three days.
  Arms: Arm 2- prophylaxis treatment

SUMMARY:
The primary objectives of the study are to evaluate the efficacy of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection (FRSW107) in the Prevention and Treatment of Bleeding in patients with hemophilia A.

The secondary objectives are to evaluate the efficacy and safety of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection (FRSW107) in the prevention and treatment of bleeding episodes, to investigate the quality of life in patients who used the FRSW107.

ELIGIBILITY:
Inclusion Criteria:

* 1)Male, aged 12 to 60 years
* 2)Severe hemophilia A. The activity of the coagulation factor VIII (FVIII:C) < 1%, and previously treated with FVIII concentrate (s) for a minimum of 150 exposure days (EDs) prior to study entry.
* 3) No history of a positive inhibitor test (< 0.6 BU) or clinical signs of decreased response to FVIII administrations within 2 years before the test or during the screening period. No Family history of inhibitors.
* 4) Non-immune deficiency, with a certain immune capacity (CD4 > 200/μL)
* 5) Platelet count > 100,000 platelets/μL.
* 6) Normal prothrombin time or INR < 1.3.
* 7) Normal previous results of vWF antigen examination.
* 8) Negative lupus anticoagulant.
* 9) the patient has a detailed record of bleeding events for at least 6 months (the subject can be admitted to the on-demand treatment group with spontaneous bleeding ≥3 times within 6 months).
* 10) Capable of understanding and willing to comply with the conditions of the protocol have read (patient and/or guardian).

Exclusion Criteria:

* 1) Hypersensitive to any of the excipients of the test materials (e.g. allergic to murine or hamster origin heterologous proteins).
* 2) History of hypersensitivity or anaphylaxis associated with any FVIII or II immunoglobulin administration.
* 3) Other coagulation disorder(s) in addition to hemophilia A.
* 4) Patients with severe heart disease, including myocardial infarction, heart failure (III or higher level).
* 5) Clinically significant of other systematic diseases: alcoholism, drug abuse, mental disorders and mental retardation.
* 6) Significant hepatic or renal impairment (ALT and AST > 2×ULN; serum bilirubin level > 3 × upper limit of normal (ULN), BUN > 2×ULN, Cr > 176.8µmol/L).
* 7) Patients who received any anticoagulant or antiplatelet therapy within one week prior screening or need to receive an anticoagulant or antiplatelet therapy during the period of clinical trials.
* 8) Patients having major surgery or receiving blood or blood components transfusion within 4 weeks prior screening or having planned major surgery schedule during the study.
* 9) Patients who previously participated in the other clinical trials within 1 month prior screening.
* 10) One or more clinically significant tests for Hepatitis B Virus Surface Antigen, Human Immunodeficiency Virus (HIV), Antisyphilitic spirulina (TPHA) and Hepatitis C Virus (HCV) Antibody.
* 11) Any life-threatening disease or condition which, according to the investigator's judgment, could not benefit from the trial participation.
* 12) Patient who is considered by the other investigators not suitable for clinical study.

NOTE:Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Hemophilia A is an X-chromosome-linked recessive inherited bleeding disorder caused by a deficiency of coagulation factor VIII (FVIII).
Enrollment: 119 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Part A - score of bleeding symptoms and Vital signs. | For the duration of study participation, 6 months.
  Response to treatment with rFVIIIFc for bleeding episodes, using the 4-point bleeding response scale.
Part B- Annualized Bleeding Rates(ABR). | For the duration of study participation, 6 months.
  Annualized bleeding rate = (number of bleeding episodes during the efficacy, period/total number of days during the efficacy period)*365.25. The efficacy period begins with the first prophylactic dose of FRSW107 and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. A bleeding episode started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. Any injection to treat the bleeding episode taken more than 72 hours after the preceding one was considered the first injection to treat a new bleeding episode at the same location. Any bleeding at a different location was considered a separate bleeding episode, regardless of time from last injection.
Part B-Number of target joints. | For the duration of study participation, 6 months.
  The joint with ≥3 times of spontaneous bleeding in 6 consecutive months is the target joint, while the joint with < 2 times of bleeding in 12 consecutive months is no longer the target joint.

SECONDARY OUTCOMES:
Part A-rFVIIIFc incremental recovery (IR). | For the duration of study participation, 6 months.
  Incremental recovery of Factor VIII (FVIII) within 1 hour after end of infusions was determined and mean recovery values were reported.
Part A -Total Dose Required for Resolution of a Bleeding Episode. | For the duration of study participation, 6 months.
  The total dose required to resolve a bleeding episode per participant, based on the efficacy period. The efficacy period begins with the first dose and ends with the last dose (for a bleed). For 'Per bleeding episode' values, for each bleeding episode, the total dose is the sum of the doses (IU/kg) administered across all injections given to treat that bleeding episode. For 'Per participant' values, the total dose (IU/kg) used to resolve each bleed is averaged across all bleeding episodes per participant.Quality of life assessment.
Part A -Number of injections required to resolve a bleeding episode. | For the duration of study participation, 6 months.
  The number of injections required to resolve a bleeding episode per participant, based on the efficacy period. The efficacy period begins with the first dose and ends with the last dose (for a bleed). All injections given from the initial sign of a bleed, until the last date/time within the bleed window are counted. The resolution of a bleed is defined as no sign of bleeding following injection for the bleed. For 'Per participant' values, the number of injections required to resolve each bleed is averaged across all bleeding episodes per participant.
Part A -Quality of life assessment. | For the duration of study participation, 6 months.
  Quality of life assessment by Haemophilia Joint Health Score（HJHS）.
Part B -Number of injections required to resolve a bleeding episode. | For the duration of study participation, 6 months.
  The number of injections required to resolve a bleeding episode per participant, based on the efficacy period. The efficacy period begins with the first prophylactic dose and ends with the last dose (for prophylaxis or a bleed). All injections given from the initial sign of a bleed, until the last date/time within the bleed window are counted. The resolution of a bleed is defined as no sign of bleeding following injection for the bleed. For 'Per participant' values, the number of injections required to resolve each bleed is averaged across all bleeding episodes per participant.
Part B -Quality of life assessment. | For the duration of study participation, 6 months.
  Quality of life assessment by Haemophilia Joint Health Score(HJHS).
Part B -Number of participants with inhibitor development | 6 months and at least 50 exposure days.
  Number of participants who developed a positive FVIII inhibitor level (≥0.6 Bethesda unit [BU]) during the study was summarized and classified as participants developing low titer inhibitor (i.e. ≤ 5.0 BU) and participants developing high titer inhibitor (i.e. > 5.0 BU).
Part B - Number of Participants With Incidence of Antibody Formation to CHINESE HAMSTER OVARY (CHO). | before and the duration of study participation, 6 months.
  A test to analyze the formation of antibodies to CHO.
Part B -Number of All Bleeds. | before and the duration of study participation, 6 months.
  The annualized number of bleeds experienced by participants.
Part B-Maximum Activity (Cmax) as Measured by the aPTT Clotting Assay | Samples taken at pre-injection, and post dose up to 96 hours at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.).
  Maximum measured concentration of rFVIIIFc.
Part B-Half-life (t½) as Measured by aPTT Clotting Assay | Samples taken at pre-injection, and post dose up to 96 hours at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.).
  Time required for the concentration of the drug to reach half of its original value.
Part B-Clearance (CL) as Measured by the aPTT Clotting Assay | Samples taken at pre-injection, and post dose up to 96 hours at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.).
  The measure of the efficiency of the body to remove the drug and the unit is the volume of the plasma or blood cleared of drug per unit time.
Part B-Volume of Distribution at Steady State (Vss) as Measured by the aPTT Clotting Assay. | Samples taken at pre-injection, and post dose up to 96 hours at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.).
  The apparent volume of distribution at steady state. (Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.).
Part B-Mean Residence Time (MRT) as Measured by the aPTT Clotting Assay. | Samples taken at pre-injection, and post dose up to 96 hours at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.).
  The average time at which the number of absorbed molecules reside in the body, after single-dose administration.
Part B-Time of Cmax (Tmax) as Measured by aPTT Clotting Assay. | Samples taken at pre-injection, and post dose up to 96 hours at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.).
  Time at which maximum activity (Cmax) is observed.
Part B-Area Under the Curve to the Last Measurable Time Point (AUClast) as Measured by aPTT Clotting Assay. | Samples taken at pre-injection, and post dose up to 96 hours at ED1 and ED35(Participants will be tested for PK assessment at timepoints throughout the study based on exposure days (ED). One ED is equivalent to a 24 hours period in which drug is dosed.).
  Area under the plasma concentration time-curve from zero to the last measured concentration.

OTHER OUTCOMES:
Part B-Response to treatment of bleeds. | the duration of study participation, 6 months.
  Participants or caregivers were asked to assess the response to treatment of bleeds as excellent, good, moderate or poor. Percentage of bleeds per assessment was summarized and reported.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events. (SAEs) as a Measure of Safety and Tolerability | the duration of study participation, 6 months.
  An AE is any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition.

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (17):
- China (17):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Capital Medical University affiliated Beijing Children's Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan provincial People's Hospital, Zhengzhou, He'nan
  - Henan Cancer Hospital, Zhengzhou, He'nan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Jinan central hospital, Ji'nan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality